CLINICAL TRIAL: NCT06081855
Title: Predictors of Aortic Root Dilatation in Tetralogy of Fallot Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Gamal Ahmed Ramadan, Principle investigator, Assiut University
Other Study IDs: Aortic Root Dilatation in TOF
Record Dates: First submitted 2023-09-27; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Congenital Heart Disease; Aortic Root Dilatation; Tetralogy of Fallot
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Repaired TOF
  Interventions: Diagnostic Test: CT
- Unrepaired TOF
  Interventions: Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: CT — Measuring aortic root diameter by CT

SUMMARY:
* To predict vulnerable patients for aortic root dilatation in TOF patients using CT as a reliable imaging modality, thus aiding early intervention, and identifying those who will require strict follow-up.
* To assess the prevalence of TOF patients who developed aortic root dilatation, and those who were complicated with dissection, AR, and aneurysm, through collecting data from a large center (Aswan Heart Centre).
* To investigate the relationship between age at repair and the diameter of aortic root.

DETAILED DESCRIPTION:
Tetralogy of Fallot (TOF) occurs in approximately 3 to 5 of every 10,000 live births and is the most common cyanotic congenital heart defect and it exhibits four main features. These features are pulmonary stenosis, right ventricular hypertrophy, overriding aorta and ventricular septal defect. Moreover, since the survival of patients with congenital heart diseases has improved significantly in recent decades, long-term complications should be monitored cautiously. One of these complications is aortic root dilatation, attributed to increased and altered flow through the overriding aorta and an uneven sharing of conotruncal tissue between the aorta and pulmonary artery, particularly in patients who have not undergone early repair.

Despite the concern that TOF patients may harbor aortopathy that can lead to aortic regurgitation, aortic aneurysms, and, potentially, aortic dissection, the scope of the problem remains uncertain. Prevalence estimates of aortic root dilatation have ranged from 15% to 87% with the use of various criteria. Moderate to severe aortic regurgitation (AR) has also been reported in up to 12.5% of adults with TOF and dilated aortic roots. The incidence of aortic dissection and surgical intervention remains unknown. Moreover, features associated with aortic dilatation are not fully understood. Therefore, correlating and predicting vulnerable patients and identifying possible risk factors for aortic root dilatation in TOF patients, will enable more cautious follow-up and earlier intervention, thus decreasing possible morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients with TOF who either underwent or have not yet had surgical correction.
* All patients with Fallot-type DORV.
* Patients should have survived until discharge and have at least one echocardiography and CT with full data related to one or more anatomic subcomponents of the aortic root, either before surgery or during follow-up, regardless of specific duration post repair.

Exclusion Criteria:

- Patients who have contraindication for conducting cardiac CT scan. For instance, dye sensitivity, pregnancy, CKD, in addition to patients who have factors that interfere with CT image quality as metallic objects within the chest (e.g. Pacemaker).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sample size was calculated using Epi- Info7. Based on aortic dilatation is found in 84.6 in follow up CT [12] With a confidence limits 5% and a confidence level of 80% the minimum patients required for this study is 77 cases.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Aortic root diameters | Throughout the study duration, about 1 year
  : Aortic root diameters at four levels:
  1. aortic annulus (AA)
  2. sinus of Valsalva (SoV)
  3. sinotubular junction (STJ)
  4. ascending aorta (AAo). AA will be measured as the inter-commissural distance in the aortic valve, SoV will be measured at the level of maximal diameter on the axial image, STJ will be measured at the level of transitional zone from STJ to AAo, and AAo will be measured at the level of the main pulmonary artery bifurcation. Aortic cross-sectional area will be calculated by π×(diameter/2)2 The largest diameters of each aortic structure as measured based on the chest CT will be re-calculated as z-scores. In our study, "significant dilatation of the aortic structures" is defined as 95% confidence interval (z-score≥2) in diameter of each aortic structures. Echocardiography will be performed to check other cardiac deformities, including AR.

SECONDARY OUTCOMES:
Aortic valve repair or surgical or transcatheter aortic valve replacement | Throughout the study duration, about 1 year
Severity of AR at latest follow-up or before the earliest aortic valve or root intervention. | Throughout the study duration, about 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amr Elbadry, MD, Study Chair — Assiut University, Faculty of Medicine

REFERENCES:
- [Background] Expert Consensus Panel:; Miller JR, Stephens EH, Goldstone AB, Glatz AC, Kane L, Van Arsdell GS, Stellin G, Barron DJ, d'Udekem Y, Benson L, Quintessenza J, Ohye RG, Talwar S, Fremes SE, Emani SM, Eghtesady P. The American Association for Thoracic Surgery (AATS) 2022 Expert Consensus Document: Management of infants and neonates with tetralogy of Fallot. J Thorac Cardiovasc Surg. 2023 Jan;165(1):221-250. doi: 10.1016/j.jtcvs.2022.07.025. Epub 2022 Oct 26. PMID 36522807
- [Background] Goldstein BH, Petit CJ, Qureshi AM, McCracken CE, Kelleman MS, Nicholson GT, Law MA, Meadows JJ, Zampi JD, Shahanavaz S, Mascio CE, Chai PJ, Romano JC, Batlivala SP, Maskatia SA, Asztalos IB, Kamsheh AM, Healan SJ, Smith JD, Ligon RA, Pettus JA, Juma S, Raulston JEB, Hock KM, Pajk AL, Eilers LF, Khan HQ, Merritt TC, Canter M, Juergensen S, Rinderknecht FA, Bauser-Heaton H, Glatz AC. Comparison of Management Strategies for Neonates With Symptomatic Tetralogy of Fallot. J Am Coll Cardiol. 2021 Mar 2;77(8):1093-1106. doi: 10.1016/j.jacc.2020.12.048. PMID 33632484
- [Background] Niwa K, Siu SC, Webb GD, Gatzoulis MA. Progressive aortic root dilatation in adults late after repair of tetralogy of Fallot. Circulation. 2002 Sep 10;106(11):1374-8. doi: 10.1161/01.cir.0000028462.88597.ad. PMID 12221055
- [Background] Mongeon FP, Gurvitz MZ, Broberg CS, Aboulhosn J, Opotowsky AR, Kay JD, Valente AM, Earing MG, Lui GK, Fernandes SM, Gersony DR, Cook SC, Ting JG, Nickolaus MJ, Landzberg MJ, Khairy P; Alliance for Adult Research in Congenital Cardiology (AARCC). Aortic root dilatation in adults with surgically repaired tetralogy of fallot: a multicenter cross-sectional study. Circulation. 2013 Jan 15;127(2):172-9. doi: 10.1161/CIRCULATIONAHA.112.129585. Epub 2012 Dec 6. PMID 23224208
- [Background] Chong WY, Wong WH, Chiu CS, Cheung YF. Aortic root dilation and aortic elastic properties in children after repair of tetralogy of Fallot. Am J Cardiol. 2006 Mar 15;97(6):905-9. doi: 10.1016/j.amjcard.2005.09.141. Epub 2006 Feb 3. PMID 16516599
- [Background] Niwa K. Aortic root dilatation in tetralogy of Fallot long-term after repair--histology of the aorta in tetralogy of Fallot: evidence of intrinsic aortopathy. Int J Cardiol. 2005 Aug 18;103(2):117-9. doi: 10.1016/j.ijcard.2004.07.002. PMID 16080967
- [Background] Rathi VK, Doyle M, Williams RB, Yamrozik J, Shannon RP, Biederman RW. Massive aortic aneurysm and dissection in repaired tetralogy of Fallot; diagnosis by cardiovascular magnetic resonance imaging. Int J Cardiol. 2005 May 11;101(1):169-70. doi: 10.1016/j.ijcard.2004.05.037. No abstract available. PMID 15860407
- [Background] Konstantinov IE, Fricke TA, d'Udekem Y, Robertson T. Aortic dissection and rupture in adolescents after tetralogy of Fallot repair. J Thorac Cardiovasc Surg. 2010 Nov;140(5):e71-3. doi: 10.1016/j.jtcvs.2010.06.045. Epub 2010 Aug 1. No abstract available. PMID 20674941
- [Background] Colan SD, McElhinney DB, Crawford EC, Keane JF, Lock JE. Validation and re-evaluation of a discriminant model predicting anatomic suitability for biventricular repair in neonates with aortic stenosis. J Am Coll Cardiol. 2006 May 2;47(9):1858-65. doi: 10.1016/j.jacc.2006.02.020. Epub 2006 Apr 17. PMID 16682313
- [Background] Gautier M, Detaint D, Fermanian C, Aegerter P, Delorme G, Arnoult F, Milleron O, Raoux F, Stheneur C, Boileau C, Vahanian A, Jondeau G. Nomograms for aortic root diameters in children using two-dimensional echocardiography. Am J Cardiol. 2010 Mar 15;105(6):888-94. doi: 10.1016/j.amjcard.2009.11.040. PMID 20211339
- [Background] Mohammed AFA, Frick M, Kerst G, Hatam N, Elgamal MF, Essa KM, Hovels-Gurich HH, Vazquez-Jimenez JF, Zayat R. Proximal Aortic Dilatation and Pulmonary Valve Replacement in Patients with Repaired Tetralogy of Fallot: Is There a Relationship? A Cardiac Magnetic Resonance Imaging Study. J Clin Med. 2021 Nov 15;10(22):5296. doi: 10.3390/jcm10225296. PMID 34830578
- [Background] Kim W, Kwak JG, Cho S, Kim WH. Ten-year follow-up of dilatation of aortic structures in Fallot-type anomalies. Pediatr Cardiol. 2023 Oct;44(7):1552-1559. doi: 10.1007/s00246-023-03225-7. Epub 2023 Jul 5. PMID 37405457